CLINICAL TRIAL: NCT04673188
Title: Predicting Factors for the Outcome of Surgical Treatment for Patellar Instability
Acronym: MPFL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Nik Žlak (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other); University of Ljubljana (Other)
Responsible Party: Sponsor-Investigator, Nik Žlak, Principal investigator, Doctor of medicine, PhD student, University Medical Centre Ljubljana
Organization: University Medical Centre Ljubljana (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KME 0120-169/2020/4
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Patellar Dislocation
Keywords: Medial patello femoral ligament; Patellar instability; Reconstruction; Predicting factors
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Reconstruction of MPFL with or without tibial tuberositas osteotomy — Reconstruction of the medial patellofemoral ligament with autologous grafts with or without osteotomy and transfer of tibial tuberosities.

SUMMARY:
The purpose of the study is:

1. to analyze the success of operative stabilization of the patellar joint with the reconstruction of the medial patellofemoral ligament (MPFL) in terms of the subjective status of the knee, the general quality of life, and physical activity
2. to study the influence of specific preoperative (demographic and anamnestic data of the patient, radiological parameters of the knee joint) and intra-operative factors (place of femoral insertion of MPFL graft, patella height, degree of damage to the cartilaginous surfaces of the knee joint) on the subjective outcome of surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* surgical intervention with MPFL reconstruction
* with or without tibial tuberosity transposition (TTT).

Exclusion Criteria:

* trochleoplasty,
* corrective knee osteotomy
* reparative cartilage treatment
* reconstruction of other knee ligaments
* meniscus repair
* movement impairments
* plegia
* paresis
* neuromuscular diseases
* participation rejection
* rejection to complete the control questionnaires
* lack of understanding of the Slovenian language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change of subjective knee status evaluated with EQ-5D | 2-8 years
  It is expected that the subjective status of the knee will significantly improve after surgical stabilisation of the patellar joint. The change in subjective knee status will be measured with EQ-5D (European quality of life in 5 dimensions; min 0, max 100). Higher scores on the questioner mean a better outcome.
Change of subjective knee status evaluated with KOOS | 2-8 years
  It is expected that the subjective status of the knee will significantly improve after surgical stabilisation of the patellar joint. The change in subjective knee status will be measured with KOOS (Knee osteoarthritis outcome score; min 0, max 100). Higher scores on the questioner mean a better outcome.
Change of subjective knee status on Tegner activity scale | 2-8 years
  It is expected that the subjective status of the knee will significantly improve after surgical stabilisation of the patellar joint. The change in subjective knee status will be measured with Tegner activity scale (min 0, max 10). Higher scores on the scale mean a better outcome.
Change of subjective knee status evaluated with Kujala score | 2-8 years
  It is expected that the subjective status of the knee will significantly improve after surgical stabilisation of the patellar joint. The change in subjective knee status will be measured with Kujala questioner (min 0, max100). Higher score means a better outcome.
Change of subjective knee status on IKDC | 2-8 years
  It is expected that the subjective status of the knee will significantly improve after surgical stabilisation of the patellar joint. The change in subjective knee status will be assessed with IKDC (International knee documentation committeemin; 0, max 100) questioner. Higher score on the questioner means a better outcome.

SECONDARY OUTCOMES:
Patellar position change | 2-8 years
  The height of the patella in the late post-operative period is not expected to differ from its position immediately after the procedure. The patellar height will be assessed with Caton-Deschamp index on standard lateral X-rays before surgery, immediately after surgery and at least six months after surgery. Reference values for normal patellar height are 0.8 - 1.2.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedic Surgery of the Ljubljana University Medical Centre, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided